CLINICAL TRIAL: NCT01166373
Title: Long-Term Effectiveness Of Sacrospinous Ligament Fixation vs Uterosacral Ligament Suspension With and Without Perioperative Behavioral Therapy/Pelvic Muscle Training: Extended Operations & Pelvic Muscle Training Of Apical Support Loss Study
Brief Title: The Extended Operations And Pelvic Muscle Training In The Management Of Apical Support Loss Study
Acronym: E-OPTIMAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NICHD Pelvic Floor Disorders Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Other
Other Study IDs: 16P01S
Record Dates: First submitted 2010-07-19; First posted 2010-07-21 (Estimated); Results first posted 2020-09-28 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Pelvic Organ Prolapse
Keywords: prolapse; urinary incontinence; uterosacral vaginal vault ligament suspension; sacrospinous ligament fixation; behavioral therapy; pelvic muscle training
MeSH Terms: conditions — Pelvic Organ Prolapse; Prolapse; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Enrollment video arm (Experimental): Arm of subjects that will be shown a standardized video detailing the importance of long-term follow-up studies for pelvic organ prolapse prior to the informed consent process.
  Interventions: Behavioral: Enrollment video
- No video intervention arm (No Intervention): This group of subjects will not view a standardized video detailing the importance of long-term follow-up studies for pelvic organ prolapse prior to the informed consent process.
- ULS (Experimental): Uterosacral Ligament Suspension was one of the randomized surgical treatments in the OPTIMAL study
  Interventions: Procedure: ULS
- SSLF (Experimental): Sacrospinous Ligament Fixation was one of the randomized surgical treatments in the OPTIMAL study.
  Interventions: Procedure: SSLF
- PMT (Experimental): Perioperative Behavioral Therapy/Pelvic Muscle Training was one of the randomized non-surgical (behavioral) interventions in the OPTIMAL study.
  Interventions: Behavioral: PMT
- Usual Care (Other): No Perioperative Behavioral Therapy/Pelvic Muscle Training (i.e., usual care) was one of the randomized non-surgical (behavioral) interventions in the OPTIMAL study.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Enrollment video — Standardized video detailing the importance of long-term follow-up studies for pelvic organ prolapse prior to the informed consent process
  Arms: Enrollment video arm
Procedure: SSLF — sacrospinous ligament fixation to suspend the vaginal apex
  Arms: SSLF
Procedure: ULS — uterosacral ligament suspension to suspend the vaginal apex
  Arms: ULS
Behavioral: PMT — perioperative behavioral therapy / pelvic muscle training with formal individualized PMT program that begins two to four weeks prior to surgery and continues for three months after surgery
  Arms: PMT
Other: Usual Care — usual care both before and after prolapse surgery with respect to pelvic muscle training
  Arms: Usual Care

SUMMARY:
Women will be invited to participate in E-OPTIMAL at their last clinical follow-up visit for OPTIMAL (at 24 months post surgery). E-OPTIMAL is an extension of the ongoing OPTIMAL study and no new study treatment interventions will be given. Rather an enrollment intervention will be investigated with potential E-OPTIMAL participants randomly assigned to watch a standardized video prior to consent or undergo the standard informed consent process. The standardized video will review the rationale for women's health research, the importance of long-term follow-up and a detailed invitation to participate in E-OPTIMAL. The video has undergone review by potential subjects, coordinators and physician researchers to ensure that the relevance and importance of issues potentially impacting on long-term participation in studies such as E-OPTIMAL are covered. Participation in E-OPTIMAL will occur up to three additional years. Women will be strongly encouraged to participate in annual examinations and annual telephone surveys but may participate in only one of these study parts if needed.

We propose to test the following null hypotheses:

1. There will be no difference in time to surgical failure between uterosacral vaginal vault ligament suspension (ULS) and sacrospinous ligament fixation (SSLF) up to 5 years after surgery.
2. The addition of a standardized video detailing the importance of long-term follow-up studies for POP to the informed consent process will not improve enrollment or retention in E-OPTIMAL.

DETAILED DESCRIPTION:
The goal of this long-term follow-up study is to extend the follow-up of women in the OPTIMAL study up to 5 years from the time of surgery and to compare the success and complication rates of the two surgical treatment groups over this extended time period. The Operations and Pelvic Muscle Training in the Management of Apical Support Loss (OPTIMAL) study is a randomized trial designed to compare sacrospinous ligament fixation (SSLF) to uterosacral vaginal vault ligament suspension (ULS) and to assess the role of perioperative behavioral therapy/pelvic muscle training (PMT) in women undergoing vaginal surgery for apical or uterine prolapse and stress urinary incontinence (SUI).

The OPTIMAL study includes a two-year follow up from the time of surgery, which is too short to evaluate the long-term sequelae of the surgical procedures. A further goal of E-OPTIMAL is to investigate a strategy for improving enrollment and retention in long-term studies of women undergoing surgery for pelvic organ prolapse and SUI, by randomizing subjects to two different recruitment methods.

The primary aims of this extension study are to compare SSLF and ULS for the following outcomes up to 5 years after surgery in women with Stage 2-4 prolapse involving the vaginal apex or uterus and stress urinary incontinence:

1. time to surgical failure;
2. the long-term functional and health-related quality of life (QOL), adjusted for PMT treatment group;
3. the annual and cumulative incidence, resolution, and persistence of pelvic floor symptoms (urinary, bowel, and prolapse), adjusted for PMT treatment group.

An additional primary aim (aim 4) is to determine whether exposure to a standardized video detailing the importance of long-term follow-up studies for pelvic organ prolapse prior to the informed consent process will improve enrollment and/or retention in E-OPTIMAL. We will utilize a conceptual framework that assesses three concepts (motivation, barriers and pragmatic issues) at two levels (study level and personal/individual level). This conceptual framework was developed following a review of the scant available literature on the topic, as well as during discussions with investigators who are experienced in recruiting and retaining participants in pelvic floor disorders studies.

ELIGIBILITY:
Inclusion Criteria:

1. Completion of the Year 2 OPTIMAL in-person visit

Exclusion Criteria:

1. Inability to provide informed consent.
2. Subjects who are long-term residents of a skilled nursing facility (that is, residency is not limited to short-term rehabilitation) at the time of enrollment into E-OPTIMAL. Note: Subjects unable to return for annual visits are not excluded as they can participate in the telephone interview. However, every attempt will be made to encourage in-person participation.

Criteria for termination of participation:

(Due to evidence or likelihood that the subject can no longer consent for herself)

1. Subjects 75 years and older that fail the telephone mini-mental status examination. If the participant gets 5 or more of the 10 items "incorrect" the interviewer says "thank you very much for your time, that completes the interview for today." In other words, the interviewer in no way implies to the participant that they did not "pass" a test to continue. The interviewer contacts the appropriate site coordinator immediately after the interview to let them know of the outcome.
2. Subjects younger than 75 who appear to have cognitive deficits during the quality of life telephone interview will be administered the mini-mental status examination; those who fail will be excluded from further participation. (Proxy respondents will not be used.) Subjects who appear to have cognitive deficits during the in-person visit or site telephone interview will be withdrawn from the study by the study coordinator.
3. Subjects who become long-term residents of a skilled nursing facility.
4. Withdrawal of consent. Verbal assent will be obtained prior to each telephone interview and each in-person visit.

Note: Subjects that are unable to complete telephone interviews (for example, because of hearing loss) may complete the interview portion of the survey in person, either at the site or in the home.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2010-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D. Barber, MD, Principal Investigator — The Cleveland Clinic; Eric Jelovsek, MD, Principal Investigator — The Cleveland Clinic
Locations (7):
- United States (7):
  - University of Alabama, Birmingham, Alabama
  - University of California, San Diego Medical Center, La Jolla, California
  - Loyola University Medical Center, Maywood, Illinois
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Texas Southwestern, Dallas, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jakus-Waldman S, Brubaker L, Jelovsek JE, Schaffer JI, Ellington DR, Mazloomdoost D, Whitworth R, Gantz MG; NICHD Pelvic Floor Disorders Network (PFDN). Risk Factors for Surgical Failure and Worsening Pelvic Floor Symptoms Within 5 Years After Vaginal Prolapse Repair. Obstet Gynecol. 2020 Nov;136(5):933-941. doi: 10.1097/AOG.0000000000004092. PMID 33030871
- [Derived] Meyer I, Whitworth RE, Lukacz ES, Smith AL, Sung VW, Visco AG, Ackenbom MF, Wai CY, Mazloomdoost D, Gantz MG, Richter HE; NICHD Pelvic Floor Disorders Network and the National Institutes of Health Office of Research on Women's Health. Outcomes of native tissue transvaginal apical approaches in women with advanced pelvic organ prolapse and stress urinary incontinence. Int Urogynecol J. 2020 Oct;31(10):2155-2164. doi: 10.1007/s00192-020-04271-y. Epub 2020 Mar 7. PMID 32146521
- [Derived] Brubaker L, Jelovsek JE, Lukacz ES, Balgobin S, Ballard A, Weidner AC, Gantz MG, Whitworth R, Mazloomdoost D; Eunice Kennedy Shriver National Institute of Child Health and Human Development Pelvic Floor Disorders Network. Recruitment and retention: A randomized controlled trial of video-enhanced versus standard consent processes within the E-OPTIMAL study. Clin Trials. 2019 Oct;16(5):481-489. doi: 10.1177/1740774519865541. Epub 2019 Jul 26. PMID 31347384
- [Derived] Jelovsek JE, Barber MD, Brubaker L, Norton P, Gantz M, Richter HE, Weidner A, Menefee S, Schaffer J, Pugh N, Meikle S; NICHD Pelvic Floor Disorders Network. Effect of Uterosacral Ligament Suspension vs Sacrospinous Ligament Fixation With or Without Perioperative Behavioral Therapy for Pelvic Organ Vaginal Prolapse on Surgical Outcomes and Prolapse Symptoms at 5 Years in the OPTIMAL Randomized Clinical Trial. JAMA. 2018 Apr 17;319(15):1554-1565. doi: 10.1001/jama.2018.2827. PMID 29677302

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The goal of the video/no video intervention was to gauge differences in recruitment for and retention in E-OPTIMAL, thus the video/no video randomization occurred before E-OPTIMAL consent.
Pre-assignment Details: Treatment groups are from the original OPTIMAL trial. Participants in the E-OPTIMAL trial were recruited from OPTIMAL participants that completed the Year 2 OPTIMAL visit.
Groups:
- SSLF+BPMT: Sacrospinous Ligament Fixation plus Perioperative Behavioral Therapy/Pelvic Muscle Training
- SSLF+USUAL: Sacrospinous Ligament Fixation plus No Perioperative Behavioral Therapy/Pelvic Muscle Training
- ULS+BPMT: Uterosacral Ligament Suspension plus Perioperative Behavioral Therapy/Pelvic Muscle Training
- ULS+USUAL: Uterosacral Ligament Suspension plus No Perioperative Behavioral Therapy/Pelvic Muscle Training
Period: Overall Study
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Started (Randomized in Primary OPTIMAL Trial) | 95 | 91 | 91 | 97
Completed OPTIMAL Year 2 Visit | 81 | 80 | 79 | 87
Randomized to Video (Prior to E-OPTIMAL consent. Used only to assess recruitment and retention regardless of treatment) | 32 | 43 | 38 | 40
Randomized to No Video (Prior to E-OPTIMAL consent. Used only to assess recruitment and retention regardless of treatment) | 45 | 30 | 34 | 42
Consented to Participate E-OPTIMAL | 72 | 66 | 69 | 78
Completed E-OPTIMAL Year 3 Visit | 70 | 66 | 66 | 77
Completed E-OPTIMAL Year 4 Visit | 67 | 61 | 63 | 68
Completed E-OPTIMAL Year 5 Visit | 62 | 56 | 62 | 64
Completed (Included in Primary Analysis) | 90 | 87 | 87 | 92
Not Completed | 5 | 4 | 4 | 5
Not completed — Lost to Follow-up | 3 | 2 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 2 | 2 | 3
Not completed — Physician Decision | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL | Total
Number analyzed (Participants) | 72 | 66 | 69 | 78 | 285
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (10.8) | 58.6 (10.6) | 58.7 (10.5) | 56.3 (11.2) | 57.2 (10.8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 72 | 66 | 69 | 78 | 285
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 2
  Asian | 0 | 2 | 0 | 0 | 2
  Black or African American | 7 | 3 | 7 | 4 | 21
  Other | 5 | 5 | 4 | 8 | 22
  White | 59 | 55 | 58 | 66 | 238
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latina | 15 | 10 | 13 | 18 | 56
  Not Hispanic/Latina | 57 | 56 | 56 | 60 | 229
Insurance: Private/HMO [Count of Participants; unit: Participants]
  No | 70 | 65 | 68 | 76 | 279
  Yes | 2 | 1 | 1 | 2 | 6
Insurance: Medicare or Medicaid [Count of Participants; unit: Participants]
  No | 55 | 46 | 47 | 56 | 204
  Yes | 17 | 20 | 22 | 22 | 81
Insurance: Self-pay [Count of Participants; unit: Participants]
  No | 70 | 65 | 68 | 76 | 279
  Yes | 2 | 1 | 1 | 2 | 6
Insurance: Other [Count of Participants; unit: Participants]
  No | 57 | 55 | 59 | 60 | 231
  Yes | 15 | 11 | 10 | 18 | 54
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.2 (6.5) | 28.2 (5.3) | 28.8 (4.9) | 28.3 (5.2) | 28.9 (5.5)
Current Smoker [Count of Participants; unit: Participants]
  No | 64 | 61 | 64 | 73 | 262
  Yes | 8 | 5 | 5 | 5 | 23
Diabetes [Count of Participants; unit: Participants]
  Unknown | 4 | 2 | 0 | 1 | 7
  No | 59 | 59 | 58 | 72 | 248
  Yes | 9 | 5 | 11 | 5 | 30
Connective tissue disease [Count of Participants; unit: Participants]
  Unknown | 1 | 1 | 0 | 3 | 5
  No | 70 | 65 | 68 | 72 | 275
  Yes | 1 | 0 | 1 | 3 | 5
Number of Vaginal Deliveries [Median (Full Range); unit: Deliveries] | 3 [0 to 8] | 2 [0 to 12] | 3 [0 to 15] | 3 [0 to 9] | 3 [0 to 15]
Number of Cesarean Deliveries [Median (Full Range); unit: Deliveries] | 0 [0 to 4] | 0 [0 to 2] | 0 [0 to 4] | 0 [0 to 2] | 0 [0 to 4]
Estrogen Use: Oral or patch [Count of Participants; unit: Participants]
  No | 63 | 56 | 60 | 70 | 249
  Yes | 9 | 10 | 9 | 8 | 36
Estrogen Use: Vaginal cream or tablets [Count of Participants; unit: Participants]
  No | 59 | 50 | 49 | 60 | 218
  Yes | 13 | 16 | 20 | 18 | 67
Menstrual Status [Count of Participants; unit: Participants]
  Not sure | 5 | 4 | 3 | 3 | 15
  Postmenopausal | 42 | 48 | 49 | 49 | 188
  premenopausal | 25 | 14 | 17 | 26 | 82
Hysterectomy [Count of Participants; unit: Participants]
  No | 58 | 42 | 52 | 59 | 211
  Yes | 14 | 24 | 17 | 19 | 74
Prior SUI Surgery [Count of Participants; unit: Participants]
  No | 71 | 62 | 67 | 75 | 275
  Yes | 1 | 4 | 2 | 3 | 10
Prior POP Surgery [Count of Participants; unit: Participants]
  No | 68 | 58 | 67 | 74 | 267
  Yes | 4 | 8 | 2 | 4 | 18
Pelvic Organ Prolapse-Q stage [Count of Participants; unit: Participants] — The POP-Q assessment is a tool that measure the severity of prolapse. It measures nine points in the vagina with the hymen being the reference point. The distance to the reference point (in cm) is measured for the prolapsed and the severity stage is calculated. Higher stages indicate worse prolapse.
  Participants
    2 | 27 | 23 | 26 | 31 | 107
    3 | 43 | 37 | 41 | 45 | 166
    4 | 2 | 6 | 2 | 2 | 12

OUTCOME MEASURES:

1. Primary Outcome: Surgical Failure
Description: Surgical failure was defined as Pelvic Organ Prolapse Quantification (POP-Q) point C descended more than one-third of total vaginal length; POPQ points Aa, Ba, Ap, or Bp were beyond the hymen; bothersome vaginal bulge symptoms were reported by the participant; or the participant received retreatment. The apex is point C (cervix), and posteriorly is point D (pouch of Douglas). In women after hysterectomy, point C is the vaginal cuff and point D is omitted. This outcome measure is cumulatively across the original OPTIMAL trial and continued through the E-OPTIMAL follow-up with non-failures tracked either until failure or until study completion/dropping out of the study (lost to follow-up, withdrawal, etc.)
Time Frame: 6 months and 1, 2, 3, 4, and 5 years
Population: The primary analysis was conducted using an intention-to-treat principle as closely as possible by analyzing all successfully followed up participants in the OPTIMAL treatment group to which they were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 90 | 87 | 87 | 92
Participants
  0.5 years: number analyzed (Participants) | 90 | 87 | 86 | 91
  0.5 years: Failure | 17 | 22 | 20 | 14
  0.5 years: Non-failure | 73 | 65 | 66 | 77
  1 years: number analyzed (Participants) | 86 | 86 | 86 | 91
  1 years: Failure | 28 | 35 | 30 | 29
  1 years: Non-failure | 58 | 51 | 56 | 62
  2 years: number analyzed (Participants) | 82 | 84 | 83 | 89
  2 years: Failure | 31 | 45 | 39 | 37
  2 years: Non-failure | 51 | 39 | 44 | 52
  3 years: number analyzed (Participants) | 76 | 78 | 77 | 81
  3 years: Failure | 37 | 52 | 46 | 41
  3 years: Non-failure | 39 | 26 | 31 | 40
  4 years: number analyzed (Participants) | 71 | 77 | 75 | 75
  4 years: Failure | 41 | 55 | 49 | 43
  4 years: Non-failure | 30 | 22 | 26 | 32
  5 years: number analyzed (Participants) | 69 | 77 | 75 | 70
  5 years: Failure | 47 | 57 | 49 | 45
  5 years: Non-failure | 22 | 20 | 26 | 25

2. Primary Outcome: Recruitment Into E-OPTIMAL
Description: Eligible OPTIMAL participants were to receive a video (or no video) about the importance of follow-up in clinical trials. The outcome is measured as the number of OPTIMAL participants that consented to participate in E-OPTIMAL.
Time Frame: At 24 Months post OPTIMAL Treatment
Population: The objective of the Outcome Measure was to compare retention rates for the "Enrollment video arm" and "No video arm", and the OPTIMAL treatment received was not relevant to this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Enrollment Video Arm | No Video Intervention Arm
Number analyzed (Participants) | 153 | 151
Participants
  Consented to E-OPTIMAL | 142 | 143
  Did not Consent to E-OPTIMAL | 11 | 8

3. Primary Outcome: Retention in E-OPTIMAL
Description: Retention is defined as those participants who consented to participate in E-OPTIMAL that remained in the E-OPTIMAL study (i.e. completed follow-up visits and were not otherwise dropped from the study).
Time Frame: 3, 4, and 5 Years Post OPTIMAL Treatment
Population: The objective of the Outcome Measure was to compare retention rates after consent into E-OPTIMAL for the "Enrollment video arm" and "No video arm", and the OPTIMAL treatment received was not relevant to this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Enrollment Video Arm | No Video Intervention Arm
Number analyzed (Participants) | 142 | 143
Participants
  3-Year Follow-up: Retained | 139 | 135
  3-Year Follow-up: Not Retained | 3 | 8
  4-Year Follow-up: Retained | 131 | 124
  4-Year Follow-up: Not Retained | 11 | 19
  5-Year Follow-up: Retained | 124 | 120
  5-Year Follow-up: Not Retained | 18 | 23

4. Secondary Outcome: Anatomic Failure
Description: Anatomic failure was defined as POPQ system point C descended more than one-third of total vaginal length; POPQ points Aa, Ba, Ap, or Bp were beyond the hymen; or the participant received retreatment during follow-up. This outcome measure is cumulative across the original OPTIMAL trial and continued through the E-OPTIMAL follow-up with non-failures tracked either until failure or until study completion/dropping out of the study (lost to follow-up, withdrawal, etc.)
Time Frame: 6 months and 1, 2, 3, 4, and 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 90 | 86 | 86 | 92
Participants
  0.5 years: number analyzed (Participants) | 90 | 86 | 85 | 91
  0.5 years: Failure | 10 | 12 | 13 | 11
  0.5 years: Non-failure | 80 | 74 | 72 | 80
  1 years: number analyzed (Participants) | 85 | 84 | 84 | 91
  1 years: Failure | 18 | 23 | 19 | 25
  1 years: Non-failure | 67 | 61 | 65 | 66
  2 years: number analyzed (Participants) | 82 | 81 | 80 | 87
  2 years: Failure | 23 | 31 | 25 | 29
  2 years: Non-failure | 59 | 50 | 55 | 58
  3 years: number analyzed (Participants) | 75 | 70 | 71 | 78
  3 years: Failure | 29 | 37 | 31 | 31
  3 years: Non-failure | 46 | 33 | 40 | 47
  4 years: number analyzed (Participants) | 69 | 69 | 68 | 71
  4 years: Failure | 33 | 40 | 32 | 33
  4 years: Non-failure | 36 | 29 | 36 | 38
  5 years: number analyzed (Participants) | 66 | 68 | 67 | 66
  5 years: Failure | 38 | 42 | 33 | 35
  5 years: Non-failure | 28 | 26 | 34 | 31

5. Secondary Outcome: Bothersome Bulge Symptoms
Description: Bothersome bulge symptoms were reported by the participant in response to the questions, 'Do you usually have a sensation of bulging or protrusion from the vaginal area?' or 'Do you usually have a bulge or something falling out that you can see or feel in the vaginal area?' on the Pelvic Floor Disorders Inventory. An answer of "Yes" to either question indicates a failure while an answer to "No" for both questions indicates a non-failure.This outcome measure is cumulative across the original OPTIMAL trial and continued through the E-OPTIMAL follow-up with non-failures tracked either until failure or until study completion/dropping out of the study (lost to follow-up, withdrawal, etc.)
Time Frame: 6 months and 1, 2, 3, 4, and 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 90 | 88 | 87 | 94
Participants
  0.5 years: number analyzed (Participants) | 90 | 85 | 84 | 93
  0.5 years: Failure | 10 | 12 | 8 | 5
  0.5 years: Non-failure | 80 | 73 | 76 | 88
  1 years: number analyzed (Participants) | 89 | 83 | 82 | 90
  1 years: Failure | 21 | 19 | 15 | 9
  1 years: Non-failure | 68 | 64 | 67 | 81
  2 years: number analyzed (Participants) | 85 | 83 | 79 | 86
  2 years: Failure | 24 | 27 | 21 | 17
  2 years: Non-failure | 61 | 56 | 58 | 69
  3 years: number analyzed (Participants) | 74 | 74 | 71 | 75
  3 years: Failure | 27 | 29 | 28 | 20
  3 years: Non-failure | 47 | 45 | 43 | 55
  4 years: number analyzed (Participants) | 72 | 72 | 70 | 68
  4 years: Failure | 27 | 32 | 31 | 22
  4 years: Non-failure | 45 | 40 | 39 | 46
  5 years: number analyzed (Participants) | 66 | 68 | 68 | 65
  5 years: Failure | 30 | 34 | 33 | 23
  5 years: Non-failure | 36 | 34 | 35 | 42

6. Secondary Outcome: Retreatment for Pelvic Organ Prolapse
Description: Retreatment is defined as any additional POP surgery or the use of pessary. This outcome measure is cumulative across the original OPTIMAL trial and continued through the E-OPTIMAL follow-up with non-retreatments tracked either until retreatment or until study completion/dropping out of the study (lost to follow-up, withdrawal, etc.)
Time Frame: 6 months and 1, 2, 3, 4, and 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 93 | 86 | 86 | 93
Participants
  0.5 years: number analyzed (Participants) | 91 | 86 | 83 | 92
  0.5 years: Retreated | 1 | 0 | 1 | 0
  0.5 years: Not retreated | 90 | 86 | 82 | 92
  1 years: number analyzed (Participants) | 85 | 85 | 81 | 89
  1 years: Retreated | 2 | 3 | 2 | 2
  1 years: Not retreated | 83 | 82 | 79 | 87
  2 years: number analyzed (Participants) | 81 | 80 | 79 | 87
  2 years: Retreated | 5 | 3 | 6 | 2
  2 years: Not retreated | 76 | 77 | 73 | 85
  3 years: number analyzed (Participants) | 68 | 62 | 65 | 70
  3 years: Retreated | 7 | 3 | 10 | 2
  3 years: Not retreated | 61 | 59 | 55 | 68
  4 years: number analyzed (Participants) | 59 | 55 | 62 | 57
  4 years: Retreated | 7 | 4 | 10 | 5
  4 years: Not retreated | 52 | 51 | 52 | 52
  5 years: number analyzed (Participants) | 60 | 54 | 61 | 59
  5 years: Retreated | 8 | 4 | 10 | 6
  5 years: Not retreated | 52 | 50 | 51 | 53

7. Other Pre Specified Outcome: Number of Participants With Granulation Tissue
Description: Cumulative number of participants with granulation tissue. Granulation tissue was reported on the adverse event log.
Time Frame: 2, 3, 4, and 5 years
Population: An analysis which included all participants that completed the primary OPTIMAL trial though 2 years and who were consented to extended follow-up through 5 years.
Measure: Count of Participants; unit: Participants
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 72 | 66 | 69 | 78
Participants
  2 years: No | 58 | 60 | 52 | 63
  2 years: Yes | 14 | 6 | 17 | 15
  3 years: number analyzed (Participants) | 68 | 60 | 65 | 71
  3 years: No | 54 | 54 | 48 | 56
  3 years: Yes | 14 | 6 | 17 | 15
  4 years: number analyzed (Participants) | 63 | 55 | 61 | 66
  4 years: No | 49 | 49 | 43 | 50
  4 years: Yes | 14 | 6 | 18 | 16
  5 years: number analyzed (Participants) | 58 | 54 | 60 | 61
  5 years: No | 43 | 48 | 41 | 45
  5 years: Yes | 15 | 6 | 19 | 16

8. Other Pre Specified Outcome: Number of Participants With Suture Exposure
Description: Cumulative number of participants with suture exposure. Suture exposure was reported on the adverse event log.
Time Frame: 2, 3, 4, and 5 years
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 72 | 66 | 69 | 78
Participants
  2 years: No | 57 | 55 | 60 | 60
  2 years: Yes | 15 | 11 | 9 | 18
  3 years: number analyzed (Participants) | 69 | 61 | 66 | 71
  3 years: No | 53 | 50 | 57 | 52
  3 years: Yes | 16 | 11 | 9 | 19
  4 years: number analyzed (Participants) | 66 | 56 | 61 | 66
  4 years: No | 49 | 44 | 51 | 46
  4 years: Yes | 17 | 12 | 10 | 20
  5 years: number analyzed (Participants) | 59 | 54 | 60 | 60
  5 years: No | 42 | 42 | 49 | 40
  5 years: Yes | 17 | 12 | 11 | 20

9. Other Pre Specified Outcome: Number of Participants With Midurethral Sling Erosion or Exposure
Description: Cumulative number of participants with mesh erosion or exposure. Mesh erosion and exposure was reported on the adverse event log.
Time Frame: 2, 3, 4, and 5 years
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 72 | 66 | 69 | 78
Participants
  2 years: number analyzed (Participants) | 71 | 66 | 69 | 78
  2 years: No | 70 | 66 | 68 | 78
  2 years: Yes | 1 | 0 | 1 | 0
  3 years: number analyzed (Participants) | 67 | 60 | 64 | 70
  3 years: No | 65 | 59 | 63 | 70
  3 years: Yes | 2 | 1 | 1 | 0
  4 years: number analyzed (Participants) | 63 | 54 | 59 | 63
  4 years: No | 60 | 53 | 58 | 63
  4 years: Yes | 3 | 1 | 1 | 0
  5 years: number analyzed (Participants) | 56 | 52 | 56 | 57
  5 years: No | 53 | 51 | 54 | 57
  5 years: Yes | 3 | 1 | 2 | 0

10. Other Pre Specified Outcome: Number of Participants With Pelvic Organ Prolapse Surgery
Description: Cumulative number of participants with pelvic organ prolapse. Pelvic organ prolapse was reported on the adverse event log.
Time Frame: 2, 3, 4, and 5 years
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 72 | 66 | 69 | 78
Participants
  2 years: No | 72 | 64 | 67 | 76
  2 years: Yes | 0 | 2 | 2 | 2
  3 years: number analyzed (Participants) | 65 | 61 | 63 | 70
  3 years: No | 64 | 59 | 58 | 68
  3 years: Yes | 1 | 2 | 5 | 2
  4 years: number analyzed (Participants) | 56 | 54 | 60 | 57
  4 years: No | 55 | 51 | 55 | 53
  4 years: Yes | 1 | 3 | 5 | 4
  5 years: number analyzed (Participants) | 57 | 53 | 59 | 59
  5 years: No | 55 | 50 | 54 | 54
  5 years: Yes | 2 | 3 | 5 | 5

11. Other Pre Specified Outcome: PGI-I
Description: The Patient Global Impression of Improvement (PGI-I) is a patient-reported measure of perceived improvement with treatment, as assessed on a scale of 1 (very much better) to 7 (very much worse).This outcome measure is shows results from the original OPTIMAL trial as well as results from the E-OPTIMAL trial (for those that consented to the extended follow-up)
Time Frame: 6 months, and 1, 2, 3, 4, and 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 72 | 66 | 69 | 78
Participants
  0.5 years: number analyzed (Participants) | 69 | 64 | 65 | 74
  0.5 years: A little better | 12 | 11 | 10 | 12
  0.5 years: A little worse | 5 | 2 | 5 | 5
  0.5 years: Much better | 23 | 22 | 17 | 20
  0.5 years: Much worse | 1 | 1 | 1 | 1
  0.5 years: No change | 2 | 1 | 2 | 3
  0.5 years: Very much better | 26 | 26 | 29 | 31
  0.5 years: Very much worse | 0 | 1 | 1 | 2
  1 years: number analyzed (Participants) | 70 | 62 | 64 | 72
  1 years: A little better | 13 | 10 | 6 | 6
  1 years: A little worse | 4 | 1 | 2 | 6
  1 years: Much better | 22 | 24 | 18 | 28
  1 years: Much worse | 0 | 0 | 1 | 0
  1 years: No change | 4 | 2 | 5 | 4
  1 years: Very much better | 26 | 25 | 30 | 27
  1 years: Very much worse | 1 | 0 | 2 | 1
  2 years: number analyzed (Participants) | 66 | 61 | 65 | 70
  2 years: A little better | 14 | 14 | 9 | 13
  2 years: A little worse | 3 | 5 | 6 | 3
  2 years: Much better | 20 | 20 | 20 | 25
  2 years: Much worse | 3 | 0 | 0 | 1
  2 years: No change | 4 | 1 | 3 | 4
  2 years: Very much better | 21 | 21 | 25 | 23
  2 years: Very much worse | 1 | 0 | 2 | 1
  3 years: number analyzed (Participants) | 64 | 60 | 60 | 68
  3 years: A little better | 5 | 19 | 10 | 13
  3 years: A little worse | 7 | 3 | 5 | 6
  3 years: Much better | 18 | 24 | 17 | 23
  3 years: Much worse | 6 | 2 | 0 | 3
  3 years: No change | 5 | 2 | 4 | 1
  3 years: Very much better | 23 | 10 | 21 | 21
  3 years: Very much worse | 0 | 0 | 3 | 1
  4 years: number analyzed (Participants) | 56 | 54 | 52 | 60
  4 years: A little better | 9 | 14 | 7 | 16
  4 years: A little worse | 4 | 6 | 1 | 2
  4 years: Much better | 21 | 19 | 14 | 19
  4 years: Much worse | 4 | 1 | 4 | 1
  4 years: No change | 3 | 2 | 4 | 2
  4 years: Very much better | 13 | 12 | 19 | 19
  4 years: Very much worse | 2 | 0 | 3 | 1
  5 years: number analyzed (Participants) | 54 | 55 | 57 | 59
  5 years: A little better | 13 | 16 | 13 | 11
  5 years: A little worse | 2 | 4 | 4 | 5
  5 years: Much better | 17 | 19 | 12 | 21
  5 years: Much worse | 4 | 0 | 6 | 2
  5 years: No change | 4 | 5 | 3 | 3
  5 years: Very much better | 12 | 11 | 18 | 15
  5 years: Very much worse | 2 | 0 | 1 | 2

12. Other Pre Specified Outcome: Change From Baseline CRAIQ Score
Description: The Pelvic Floor Impact Questionnaire measuring the impact of bladder, bowel, and vaginal symptoms on a woman's daily activities, relationships and emotions is composed of 3 scales: the Urinary Impact Questionnaire (UIQ; 4 subscales, range 0-400), the Pelvic Organ Prolapse Impact Questionnaire (POPIQ; 4 subscales, range 0-400), and the Colorectal-Anal Impact Questionnaire (CRAIQ; 4 subscales, range 0-400). Scores are calculated by multiplying the mean value of all answered questions for a subscale by 100 divided by 3. The subscales are then added together. The range of responses is: 0-400 with 0 (least negative impact) to 400 (most negative impact). Change = (Year [0.5, 1, 2, 3, 4, 5] Score - Baseline Score). Lower scores indicate better function / fewer symptoms.
Time Frame: 6 months, and 1, 2, 3, 4, and 5 years
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 66 | 60 | 62 | 74
units on a scale
  0.5 years: number analyzed (Participants) | 61 | 57 | 59 | 67
  0.5 years | -71.3 [-95.5 to -47.1] | -45.5 [-65.8 to -25.2] | -35 [-55.6 to -14.4] | -66.8 [-89.3 to -44.3]
  1 years: number analyzed (Participants) | 63 | 54 | 56 | 66
  1 years | -73.3 [-98.3 to -48.3] | -43.4 [-63.1 to -23.7] | -37.6 [-63.5 to -11.7] | -60.5 [-83.4 to -37.6]
  2 years: number analyzed (Participants) | 58 | 54 | 58 | 67
  2 years | -47.5 [-77.7 to -17.3] | -25.1 [-49 to -1.2] | -19.2 [-45.8 to 7.4] | -38.9 [-57.7 to -20.1]
  3 years: number analyzed (Participants) | 59 | 54 | 53 | 62
  3 years | -54.6 [-81.7 to -27.5] | -20.9 [-38.2 to -3.5] | -12.9 [-39.3 to 13.5] | -36.1 [-56.7 to -15.6]
  4 years: number analyzed (Participants) | 49 | 47 | 48 | 57
  4 years | -40 [-71.7 to -8.2] | -16.6 [-42.4 to 9.2] | -8.5 [-39.7 to 22.7] | -39.1 [-61.1 to -17]
  5 years: number analyzed (Participants) | 50 | 49 | 53 | 56
  5 years | -35.7 [-62.9 to -8.5] | -14.8 [-39.2 to 9.7] | 7.4 [-21.8 to 36.5] | -22.7 [-51 to 5.7]

13. Other Pre Specified Outcome: Change From Baseline POPIQ Score
Description: as for outcome 12
Time Frame: 6 months, and 1, 2, 3, 4, and 5 years
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 66 | 60 | 62 | 74
units on a scale
  0.5 years: number analyzed (Participants) | 61 | 57 | 59 | 67
  0.5 years | -95 [-123.3 to -66.7] | -61.3 [-85.6 to -37] | -55.2 [-79.5 to -30.9] | -98.6 [-122.9 to -74.4]
  1 years: number analyzed (Participants) | 63 | 54 | 56 | 66
  1 years | -100.2 [-130.5 to -70] | -68.8 [-91 to -46.6] | -58.9 [-86 to -31.8] | -95.9 [-122.1 to -69.7]
  2 years: number analyzed (Participants) | 58 | 54 | 58 | 67
  2 years | -68.9 [-102.5 to -35.3] | -56.6 [-77.9 to -35.3] | -42.8 [-71.1 to -14.4] | -79.3 [-101.4 to -57.2]
  3 years: number analyzed (Participants) | 59 | 54 | 53 | 62
  3 years | -82.6 [-112 to -53.2] | -48.7 [-66.6 to -30.8] | -29.3 [-57.3 to -1.3] | -76.9 [-99.2 to -54.6]
  4 years: number analyzed (Participants) | 49 | 47 | 48 | 57
  4 years | -84.5 [-121.8 to -47.2] | -42.3 [-64.1 to -20.6] | -32.9 [-61.7 to -4.1] | -73 [-98.6 to -47.5]
  5 years: number analyzed (Participants) | 50 | 49 | 53 | 56
  5 years | -72.1 [-103.2 to -41.1] | -50.3 [-71.8 to -28.8] | -16.8 [-43.7 to 10.2] | -71.9 [-98.2 to -45.5]

14. Other Pre Specified Outcome: Change From Baseline UIQ Score
Description: as for outcome 12
Time Frame: 6 months, and 1, 2, 3, 4, and 5 years
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 66 | 60 | 62 | 74
units on a scale
  0.5 years: number analyzed (Participants) | 61 | 57 | 59 | 67
  0.5 years | -107.7 [-133.9 to -81.6] | -85.4 [-108.7 to -62.1] | -77.3 [-102.1 to -52.4] | -116.4 [-138.6 to -94.2]
  1 years: number analyzed (Participants) | 63 | 54 | 56 | 66
  1 years | -116.3 [-143.3 to -89.3] | -92 [-113 to -71] | -84.3 [-110.2 to -58.3] | -121.8 [-146.2 to -97.4]
  2 years: number analyzed (Participants) | 58 | 54 | 58 | 67
  2 years | -90.3 [-122.8 to -57.8] | -80.4 [-102.1 to -58.6] | -67.7 [-95.7 to -39.8] | -99.1 [-121.4 to -76.8]
  3 years: number analyzed (Participants) | 59 | 54 | 53 | 62
  3 years | -94.3 [-120.7 to -67.9] | -69.1 [-87.6 to -50.7] | -59 [-84 to -34] | -92.3 [-116.4 to -68.2]
  4 years: number analyzed (Participants) | 49 | 47 | 48 | 57
  4 years | -89.5 [-124.7 to -54.3] | -68.3 [-89.8 to -46.7] | -59.2 [-87 to -31.3] | -90.3 [-117.2 to -63.4]
  5 years: number analyzed (Participants) | 50 | 49 | 53 | 56
  5 years | -75.9 [-106 to -45.7] | -72.1 [-95.2 to -49] | -47.8 [-74 to -21.7] | -84.8 [-113 to -56.6]

15. Other Pre Specified Outcome: Change From Baseline CRADI Score
Description: The Pelvic Floor Distress Inventory is a validated, self-reported instrument used to evaluate pelvic floor symptoms. It consists of 3 scales: 1. Pelvic Organ Prolapse Distress Inventory (with 3 subscales), 2. Colorectal Anal Distress Inventory (with 4 subscales), and 3. Urinary Distress Inventory (with 3 subscales). Scores are calculated by multiplying the mean value of all questions answered by 25 for the subscales and then adding the subscales. The range of responses for the CRADI is: 0-400 with 0 (least distress) to 400 (most distress). Change = (Year [0.5, 1, 2, 3, 4, 5] Score - Baseline Score). Lower scores indicate better function / fewer symptoms.
Time Frame: 6 months, and 1, 2, 3, 4, and 5 years
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 70 | 64 | 64 | 74
units on a scale
  0.5 years: number analyzed (Participants) | 67 | 62 | 61 | 71
  0.5 years | -72.3 [-88.2 to -56.4] | -71.8 [-88.7 to -54.8] | -69.6 [-87.8 to -51.4] | -56.3 [-73.7 to -38.9]
  1 years: number analyzed (Participants) | 68 | 60 | 59 | 69
  1 years | -64.1 [-81 to -47.2] | -67.5 [-85.6 to -49.5] | -77.7 [-95.7 to -59.7] | -63.3 [-81.3 to -45.4]
  2 years: number analyzed (Participants) | 63 | 58 | 60 | 69
  2 years | -46.2 [-68.8 to -23.6] | -49.1 [-70.5 to -27.6] | -62 [-81.3 to -42.8] | -50.4 [-68.9 to -31.8]
  3 years: number analyzed (Participants) | 61 | 56 | 55 | 60
  3 years | -45.3 [-68.4 to -22.2] | -53.1 [-73.6 to -32.6] | -48.7 [-69.1 to -28.3] | -44.7 [-63.4 to -26.1]
  4 years: number analyzed (Participants) | 54 | 52 | 48 | 56
  4 years | -35.1 [-58 to -12.2] | -54.1 [-75.8 to -32.3] | -44.8 [-69.6 to -19.9] | -48.8 [-71.2 to -26.4]
  5 years: number analyzed (Participants) | 51 | 52 | 55 | 57
  5 years | -37.4 [-61.1 to -13.7] | -43.1 [-61 to -25.2] | -39.1 [-60.5 to -17.6] | -39.8 [-58.7 to -20.9]

16. Other Pre Specified Outcome: Change From Baseline POPDI Score
Description: The Pelvic Floor Distress Inventory is a validated, self-reported instrument used to evaluate pelvic floor symptoms. It consists of 3 scales: 1. Pelvic Organ Prolapse Distress Inventory (with 3 subscales), 2. Colorectal Anal Distress Inventory (with 4 subscales), and 3. Urinary Distress Inventory (with 3 subscales). Scores are calculated by multiplying the mean value of all questions answered by 25 for the subscales and then adding the subscales. The range of POPDI responses is: 0-300 with 0 (least distress) to 300 (most distress). Change = (Year [0.5, 1, 2, 3, 4, 5] Score - Baseline Score). Lower scores indicate better function / fewer symptoms.
Time Frame: 6 months, and 1, 2, 3, 4, and 5 years
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 70 | 64 | 64 | 74
units on a scale
  0.5 years: number analyzed (Participants) | 67 | 62 | 60 | 71
  0.5 years | -95.1 [-108.9 to -81.4] | -90.2 [-106.3 to -74.1] | -92.3 [-110.5 to -74.1] | -72.6 [-88.3 to -57]
  1 years: number analyzed (Participants) | 68 | 60 | 59 | 69
  1 years | -90.6 [-106 to -75.2] | -96 [-112.6 to -79.5] | -91.9 [-110.7 to -73.1] | -81.1 [-93.7 to -68.4]
  2 years: number analyzed (Participants) | 63 | 59 | 60 | 69
  2 years | -76 [-94.5 to -57.5] | -79.1 [-97.2 to -61.1] | -76.9 [-96.2 to -57.7] | -65.9 [-80.5 to -51.2]
  3 years: number analyzed (Participants) | 62 | 58 | 55 | 61
  3 years | -69.5 [-86.2 to -52.8] | -77.7 [-93.9 to -61.6] | -66.9 [-87.3 to -46.5] | -61.7 [-77.6 to -45.9]
  4 years: number analyzed (Participants) | 54 | 48 | 48 | 56
  4 years | -70.7 [-87.3 to -54.1] | -78.3 [-97.8 to -58.8] | -65.1 [-88.4 to -41.9] | -62.8 [-79.5 to -46.1]
  5 years: number analyzed (Participants) | 51 | 53 | 55 | 57
  5 years | -64.8 [-83.7 to -45.9] | -75.8 [-91.9 to -59.6] | -63.7 [-82.3 to -45.1] | -61.1 [-76.6 to -45.5]

17. Other Pre Specified Outcome: Change From Baseline UDI Score
Description: The Pelvic Floor Distress Inventory is a validated, self-reported instrument used to evaluate pelvic floor symptoms. It consists of 3 scales: 1. Pelvic Organ Prolapse Distress Inventory (with 3 subscales), 2. Colorectal Anal Distress Inventory (with 4 subscales), and 3. Urinary Distress Inventory (with 3 subscales). Scores are calculated by multiplying the mean value of all questions answered by 25 for the subscales and then adding the subscales. The range of UDI responses is: 0-300 with 0 (least distress) to 300 (most distress). Change = (Year [0.5, 1, 2, 3, 4, 5] Score - Baseline Score). Lower scores indicate better function / fewer symptoms.
Time Frame: 6 months, and 1, 2, 3, 4, and 5 years
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 70 | 64 | 64 | 74
units on a scale
  0.5 years: number analyzed (Participants) | 67 | 62 | 60 | 71
  0.5 years | -105.7 [-119.3 to -92.2] | -96 [-110 to -82] | -95 [-109.9 to -80.2] | -88.9 [-103.4 to -74.4]
  1 years: number analyzed (Participants) | 67 | 60 | 59 | 69
  1 years | -102.9 [-118.4 to -87.4] | -95.9 [-110.9 to -80.8] | -94 [-110.3 to -77.7] | -96.8 [-111.3 to -82.3]
  2 years: number analyzed (Participants) | 63 | 58 | 59 | 69
  2 years | -90.8 [-109 to -72.6] | -89.1 [-104 to -74.2] | -81.2 [-98.6 to -63.9] | -81.3 [-95.4 to -67.2]
  3 years: number analyzed (Participants) | 60 | 54 | 54 | 60
  3 years | -84.9 [-102 to -67.8] | -75 [-90.3 to -59.7] | -70.5 [-88.2 to -52.8] | -72 [-87.6 to -56.5]
  4 years: number analyzed (Participants) | 53 | 46 | 48 | 54
  4 years | -81.7 [-101.9 to -61.6] | -76.2 [-93.2 to -59.2] | -70.8 [-89.5 to -52.1] | -75.3 [-91.2 to -59.5]
  5 years: number analyzed (Participants) | 50 | 51 | 53 | 57
  5 years | -73.9 [-93.3 to -54.6] | -77.9 [-94.2 to -61.5] | -69 [-85.4 to -52.7] | -74.4 [-90.1 to -58.7]

18. Other Pre Specified Outcome: Change From Baseline Hunskaar Score
Description: The Hunskaar Urinary Incontinence assessment measures the severity of a participant's urinary incontinence. Scores range from 1 to 8 with higher score indicating more severe incontinence. Change = (Year [0.5, 1, 2, 3, 4, 5] Score - Baseline Score).
Time Frame: 6 months, and 1, 2, 3, 4, and 5 years
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 69 | 64 | 64 | 74
units on a scale
  0.5 years: number analyzed (Participants) | 66 | 62 | 60 | 71
  0.5 years | -3.6 [-4.3 to -2.8] | -2.9 [-3.9 to -2] | -3.2 [-4.3 to -2.2] | -3.5 [-4.5 to -2.6]
  1 years: number analyzed (Participants) | 67 | 60 | 58 | 68
  1 years | -3.6 [-4.5 to -2.6] | -3.3 [-4.2 to -2.4] | -3.4 [-4.5 to -2.4] | -3.2 [-4.1 to -2.3]
  2 years: number analyzed (Participants) | 63 | 57 | 60 | 69
  2 years | -3 [-4.1 to -2] | -3.2 [-4.1 to -2.2] | -2.8 [-3.8 to -1.8] | -2.7 [-3.7 to -1.8]
  3 years: number analyzed (Participants) | 61 | 56 | 55 | 61
  3 years | -2.5 [-3.5 to -1.5] | -2.6 [-3.3 to -1.9] | -2.5 [-3.6 to -1.4] | -2.8 [-3.8 to -1.9]
  4 years: number analyzed (Participants) | 50 | 52 | 49 | 55
  4 years | -2.5 [-3.4 to -1.6] | -2.5 [-3.4 to -1.6] | -2.4 [-3.7 to -1.1] | -2.6 [-3.6 to -1.6]
  5 years: number analyzed (Participants) | 52 | 51 | 55 | 57
  5 years | -1.6 [-2.8 to -0.4] | -2.6 [-3.4 to -1.8] | -2 [-3.2 to -0.7] | -2.4 [-3.5 to -1.3]

19. Other Pre Specified Outcome: Change From Baseline SF-36 Physical Health Score
Description: The health assessment questionnaire Short Form 36 Version (SF-36) determines participants' overall quality of life by assessing 1. limitations in physical functioning due to health problems; 2. limitations in usual role because of physical health problems; 3. bodily pain; 4. general health perceptions; 5. vitality; 6. limitations in social functioning because of physical or emotional problems; 7. limitations in usual role due to emotional problems; and 8. general mental health. Items 1-4 primarily contribute to the physical component summary score (PCS) of the SF-36. Items 5-8 primarily contribute to the mental component summary score (MCS) of the SF-36. Scores on each item are summed and averaged (range = 0 "worst" - 100 "best"). Change = (Year [0.5, 1, 2, 3, 4, 5] Score - Baseline Score).
Time Frame: 6 months, and 1, 2, 3, 4, and 5 years
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 72 | 62 | 67 | 76
units on a scale
  0.5 years: number analyzed (Participants) | 69 | 59 | 66 | 74
  0.5 years | 7.1 [4.9 to 9.3] | 4.3 [1.4 to 7.2] | 5.6 [3.4 to 7.7] | 7.7 [5.6 to 9.7]
  1 years: number analyzed (Participants) | 65 | 58 | 63 | 71
  1 years | 8 [5.5 to 10.5] | 5.6 [2.8 to 8.3] | 6.6 [3.9 to 9.3] | 6.8 [4.2 to 9.5]
  2 years: number analyzed (Participants) | 72 | 61 | 65 | 73
  2 years | 7.6 [5 to 10.3] | 5.2 [2.6 to 7.8] | 4.9 [2.9 to 6.9] | 6.1 [4.1 to 8.1]
  3 years: number analyzed (Participants) | 64 | 56 | 58 | 65
  3 years | 4.3 [1.8 to 6.9] | 1.1 [-1.8 to 4] | 3.5 [1 to 6] | 3.1 [0.5 to 5.7]
  4 years: number analyzed (Participants) | 56 | 50 | 52 | 58
  4 years | 4.8 [2 to 7.6] | 0.3 [-2.9 to 3.5] | 2.9 [0 to 5.7] | 2.9 [0.1 to 5.6]
  5 years: number analyzed (Participants) | 54 | 50 | 55 | 57
  5 years | 3.2 [0.5 to 5.9] | 0.9 [-2.1 to 3.8] | 2.5 [-0.2 to 5.1] | 2.7 [0.2 to 5.2]

20. Other Pre Specified Outcome: Change From Baseline SF-36 Mental Health Score
Description: as for outcome 19
Time Frame: 6 months, and 1, 2, 3, 4, and 5 years
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 72 | 62 | 67 | 76
units on a scale
  0.5 years: number analyzed (Participants) | 69 | 59 | 66 | 74
  0.5 years | 2.5 [0 to 5] | 3.1 [0.5 to 5.8] | 2.6 [0.1 to 5.2] | 1.3 [-1.6 to 4.2]
  1 years: number analyzed (Participants) | 65 | 58 | 63 | 71
  1 years | 4.1 [1.5 to 6.7] | 3.4 [0.9 to 6] | 0.6 [-2.4 to 3.6] | 2.7 [-0.6 to 5.9]
  2 years: number analyzed (Participants) | 72 | 61 | 65 | 73
  2 years | 0.8 [-2 to 3.7] | 2 [-0.5 to 4.4] | 3.1 [0.7 to 5.5] | 1.6 [-1.2 to 4.5]
  3 years: number analyzed (Participants) | 64 | 56 | 58 | 65
  3 years | 3 [0 to 6] | 2.4 [-0.9 to 5.8] | 1.6 [-1.3 to 4.5] | 2.3 [-0.9 to 5.5]
  4 years: number analyzed (Participants) | 56 | 50 | 52 | 58
  4 years | 1.4 [-1.2 to 4.1] | 1.7 [-1.3 to 4.6] | 0.5 [-2.2 to 3.1] | 1.2 [-2 to 4.5]
  5 years: number analyzed (Participants) | 54 | 50 | 55 | 57
  5 years | 3.1 [-0.3 to 6.4] | 1.8 [-2 to 5.5] | 0.8 [-1.9 to 3.4] | 1.2 [-2 to 4.4]

21. Other Pre Specified Outcome: Change From Baseline Brink Score
Description: The Brink scale considers three pelvic floor muscle contraction variables: vaginal pressure or muscle force, elevation or vertical displacement of the examiner fingers, and duration of contraction. The score ranges from 3 to 12 with higher scores indicating greater PFM function. Change = (Year [0.5, 2, 3, 4, 5] Score - Baseline Score).
Time Frame: 6 months, and 2, 3, 4, and 5 years
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 68 | 64 | 68 | 76
units on a scale
  0.5 years: number analyzed (Participants) | 65 | 63 | 67 | 69
  0.5 years | 0.2 [-0.3 to 0.8] | 0 [-0.5 to 0.5] | 0.6 [0.1 to 1.1] | 0.4 [-0.1 to 0.9]
  2 years: number analyzed (Participants) | 68 | 64 | 67 | 76
  2 years | -0.1 [-0.6 to 0.4] | 0.1 [-0.5 to 0.6] | 0.4 [0 to 0.8] | 0 [-0.4 to 0.5]
  3 years: number analyzed (Participants) | 61 | 58 | 57 | 66
  3 years | 0 [-0.6 to 0.6] | -0.3 [-1 to 0.4] | 0.3 [-0.2 to 0.8] | -0.5 [-1 to 0.1]
  4 years: number analyzed (Participants) | 50 | 48 | 55 | 55
  4 years | 0.1 [-0.5 to 0.8] | -0.5 [-1.1 to 0.2] | 0.2 [-0.3 to 0.8] | -0.5 [-1.1 to 0.1]
  5 years: number analyzed (Participants) | 54 | 50 | 55 | 55
  5 years | 0.2 [-0.5 to 0.9] | -0.6 [-1.3 to 0.1] | 0.4 [-0.2 to 1] | -0.3 [-0.9 to 0.3]

22. Other Pre Specified Outcome: POP-Q Point Ba
Description: POPQ Point Ba represents the most distal (i.e. most dependent) position of any part of the upper anterior vaginal wall (between the vaginal cuff or anterior vaginal fornix and Point Aa). The range for point Ba is -3 to total vaginal length (TVL). Point Ba coincides with Point Aa (-3 cm) in a woman who has no anterior POP. In a woman with severe POP, Ba coincides with Point C. For Point Ba, better vaginal support is assigned a negative value (ie, if there is no prolapse, point Ba is -3 cm by definition). Vaginal prolapse beyond the hymen, indicating worse vaginal support, is assigned a positive value (this may be equal to the total vaginal length at the maximum).
Time Frame: 6 months, and 1, 2, 3, 4, and 5 years
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 72 | 66 | 69 | 78
cm
  0.5 years: number analyzed (Participants) | 68 | 65 | 68 | 71
  0.5 years | -1.2 [-1.5 to -0.9] | -1.2 [-1.5 to -0.9] | -1.4 [-1.7 to -1] | -1.3 [-1.6 to -1]
  1 years: number analyzed (Participants) | 66 | 63 | 66 | 72
  1 years | -0.9 [-1.3 to -0.5] | -1.2 [-1.6 to -0.8] | -1 [-1.3 to -0.7] | -1.2 [-1.5 to -0.9]
  2 years: number analyzed (Participants) | 72 | 66 | 69 | 77
  2 years | -0.9 [-1.2 to -0.5] | -0.8 [-1.1 to -0.6] | -1.1 [-1.5 to -0.8] | -1.1 [-1.4 to -0.8]
  3 years: number analyzed (Participants) | 64 | 59 | 59 | 66
  3 years | -1.1 [-1.4 to -0.7] | -0.7 [-1.1 to -0.4] | -0.8 [-1.2 to -0.4] | -1.1 [-1.4 to -0.7]
  4 years: number analyzed (Participants) | 53 | 51 | 56 | 56
  4 years | -0.8 [-1.2 to -0.3] | -0.9 [-1.3 to -0.6] | -0.8 [-1.3 to -0.3] | -1.1 [-1.5 to -0.7]
  5 years: number analyzed (Participants) | 56 | 52 | 56 | 57
  5 years | -0.8 [-1.2 to -0.3] | -1 [-1.3 to -0.6] | -0.7 [-1.2 to -0.2] | -0.9 [-1.3 to -0.4]

23. Other Pre Specified Outcome: POP-Q Point Bp
Description: POP-Q Point Bp represents the most distal position of any part of the upper posterior vaginal wall (between the vaginal cuff or posterior vaginal fornix and Point Ap). It ranges from -3 to total vaginal length (TVL). Negative values indicate vaginal support above the hymen, so the more negative number the closer to normal/perfect support; positive values show prolapse beyond the hymen, so larger positive numbers are worse prolapse.
Time Frame: 6 months, and 1, 2, 3, 4, and 5 years
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 72 | 66 | 69 | 78
cm
  0.5 years: number analyzed (Participants) | 68 | 65 | 68 | 71
  0.5 years | -2.3 [-2.5 to -2] | -2.5 [-2.7 to -2.3] | -2.2 [-2.5 to -2] | -2.2 [-2.4 to -1.9]
  1 years: number analyzed (Participants) | 66 | 63 | 66 | 72
  1 years | -2.2 [-2.4 to -2] | -2.4 [-2.6 to -2.2] | -2.2 [-2.4 to -2] | -2.2 [-2.5 to -2]
  2 years: number analyzed (Participants) | 72 | 66 | 69 | 77
  2 years | -2 [-2.2 to -1.7] | -2.3 [-2.5 to -2.1] | -2.2 [-2.4 to -2] | -2 [-2.3 to -1.8]
  3 years: number analyzed (Participants) | 64 | 59 | 59 | 66
  3 years | -2.3 [-2.5 to -2] | -2.4 [-2.6 to -2.2] | -2.1 [-2.3 to -1.9] | -2.2 [-2.5 to -1.9]
  4 years: number analyzed (Participants) | 53 | 51 | 56 | 56
  4 years | -2.2 [-2.4 to -1.9] | -2.3 [-2.5 to -2.1] | -2.2 [-2.4 to -1.9] | -2 [-2.3 to -1.7]
  5 years: number analyzed (Participants) | 56 | 52 | 56 | 57
  5 years | -2.2 [-2.4 to -2] | -2.3 [-2.5 to -2.1] | -1.9 [-2.4 to -1.4] | -1.9 [-2.2 to -1.6]

24. Other Pre Specified Outcome: POP-Q Point C
Description: POP-Q Point C is measured in cm relative to the hymen with negative values being proximal to the hymen and positive values distal to the hymen. Point C represents either the most distal edge of the cervix or the leading edge of the vaginal cuff after total hysterectomy. It ranges from -TVL to +TVL. Negative values indicate vaginal support above the hymen, so the more negative number the closer to normal/perfect support; positive values show prolapse beyond the hymen, so larger positive numbers are worse prolapse.
Time Frame: 6 months, and 1 2, 3, 4, and 5 years
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
Number analyzed (Participants) | 72 | 66 | 69 | 78
cm
  0.5 years: number analyzed (Participants) | 68 | 64 | 67 | 71
  0.5 years | -7.2 [-7.5 to -6.9] | -7.3 [-7.7 to -7] | -6.5 [-7.3 to -5.7] | -7 [-7.4 to -6.7]
  1 years: number analyzed (Participants) | 66 | 63 | 66 | 72
  1 years | -7 [-7.5 to -6.5] | -6.5 [-7.2 to -5.8] | -6.6 [-7 to -6.2] | -6.8 [-7.2 to -6.3]
  2 years: number analyzed (Participants) | 72 | 65 | 69 | 77
  2 years | -6.8 [-7.3 to -6.3] | -6.6 [-6.9 to -6.2] | -6.5 [-6.9 to -6] | -6.8 [-7.1 to -6.5]
  3 years: number analyzed (Participants) | 64 | 59 | 59 | 66
  3 years | -6.9 [-7.2 to -6.5] | -6.4 [-6.7 to -6.1] | -6.3 [-6.9 to -5.8] | -6.3 [-6.6 to -5.9]
  4 years: number analyzed (Participants) | 53 | 51 | 56 | 56
  4 years | -6.3 [-6.7 to -5.9] | -6.2 [-6.5 to -5.8] | -6.4 [-7 to -5.8] | -6.6 [-7 to -6.2]
  5 years: number analyzed (Participants) | 56 | 52 | 56 | 57
  5 years | -6.5 [-7.1 to -6] | -6.4 [-6.8 to -6] | -5.8 [-6.5 to -5.1] | -6.6 [-7.1 to -6.2]

ADVERSE EVENTS:
Time Frame: 2 years through 5 years.
Description: Only specific adverse events were recorded during the extended follow-up of the OPTIMAL trial (E-OPTIMAL). Video/No video randomization arms were only assessed with regard to retention/recruitment rates and were not expected to impact outcomes or adverse events. Adverse Events were only collected with respect to the OPTIMAL treatment received.
Arm/Group | SSLF+BPMT | SSLF+USUAL | ULS+BPMT | ULS+USUAL
All-Cause Mortality (participants affected / at risk) | 1/72 | 0/66 | 2/69 | 1/78
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/66 | 0/69 | 0/78
Other Adverse Events (participants affected / at risk) | 29/72 | 17/66 | 27/69 | 34/78
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SSLF+BPMT (N=72) | SSLF+USUAL (N=66) | ULS+BPMT (N=69) | ULS+USUAL (N=78)
Granulation tissue (Skin and subcutaneous tissue disorders) | 15 | 6 | 19 | 16
Suture exposure (Injury, poisoning and procedural complications) | 17 | 12 | 11 | 20
Midurethral sling erosion and exposure (Injury, poisoning and procedural complications) | 3 | 1 | 2 | 0
Pelvic organ prolapse surgery (Surgical and medical procedures) | 2 | 3 | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No